CLINICAL TRIAL: NCT03433885
Title: Progression of Dry Age-related Macular Degeneration (AMD): Association With Macular Pigment Optical Density (MPOD)
Brief Title: Wenzhou Dry Age-related Macular Degeneration (AMD) Progression Study
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: The Eye Hospital of Wenzhou Medical University (Other)
Responsible Party: Principal Investigator, Xiaoling Liu, Chief in retina center, The Eye Hospital of Wenzhou Medical University
Other Study IDs: kyk20175
Record Dates: First submitted 2018-01-30; First posted 2018-02-15 (Actual); Last update posted 2021-02-24 (Actual); Status verified 2021-02

CONDITIONS: Macular Pigment Optical Density
Keywords: macular pigment optical density (MPOD); Age-related Macular Degeneration (AMD); drusen; Chroidal neovascularization (CNV); lutein; zeaxanthin
MeSH Terms: conditions — Macular Degeneration

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Progressors: Progressors are those individuals with early or intermediate AMD at baseline who progress to advanced AMD during follow-up, and individuals with advanced AMD in one eye at baseline who progress to advanced AMD in both eyes.
- Nonprogressor: Nonprogressors are those individuals with early or intermediate AMD at baseline who do not progressed to advanced AMD during follow-up, and individuals with advanced AMD in one eye at baseline who do not progress to advanced AMD in fellow eye.

SUMMARY:
To evaluate the correlation between macular pigment optical density (MPOD) levels and risk of progression in patients with age-related macular degeneration

DETAILED DESCRIPTION:
Age-related macular degeneration (AMD) is the leading cause of blindness in the elderly.[1] The disease is categorized into early, intermediate, or advanced stages based on the severity of symptoms. The advanced stage, including GA and CNV, involves central region of the retina, which leads to a gradual or rapid loss of photoreceptors and central vision.

The macular pigment (MP) consists of xanthophyll, which is formed from the yellow carotenoid lutein, zeaxanthin, and meso-zeaxanthin.These pigments play an important role in protecting the retina against oxidative stress through different mechanisms[6]. Many studies have shown a various association of AMD and MP.Blue Mountain Eye Study revealed low dietary intake of lutein and zeaxanthin is associated with a higher risk of AMD. However, dry and wet subtypes of AMD may have different etiologies and risk factors. Little is known whether longitudinal study of macular pigment optical density (MPOD) is related to AMD progression.

A comprehensive ophthalmologic examination including fundus photography,OCT and MPOD was performed at baseline, and semiannually thereafter for 3 years. Fundus reflectance (VISUCAM 500, reflectance of a single 460 nm wavelength) was used to measure the MPOD levels. Associated risk factors including body-mass index (BMI), smoking, diet, and cardiovascular diseases were documented. Drusen characteristics (size, type, area), pigmentary abnormalities (increased pigment, depigmentation, geographic atrophy), and presence of abnormalities characteristic of neovascular AMD were graded. For estimations of AMD progression , a 9-step severity scale that combines a 6-step drusen area scale with a 5-step pigmentary abnormality scale is used.

In this study, we are going to investigate a 3-year study of incidence and progression for AMD and associated risk factors, in a population-based cohort of Chinese aged 45 years and older living in the city of Wenzhou.

ELIGIBILITY:
Inclusion Criteria:

* subject is diagnosed with either CNV, dry AMD
* 45 years of age or older
* provides signed and dated informed consent

Exclusion Criteria:

* Ocular condition in the study eye which may impact vision and confound study outcomes
* Presence of macular edema like retinal vascular diseases or diabetic retinopathy
* active inflammation ofr infection in the study eye
* high myopia（ ≥6D ）

Min Age: 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Chinese subjects aged 45 years and older living in the city of Wenzhou diagnosed with either CNV or dry AMD
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2018-01-01 (Actual); Primary Completion 2021-12-31 (Estimated); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
Association between changes of macular pigment optical density (MPOD) level and incidence rates of advanced AMD | from baseline to month 36
  Incident advanced AMD was evaluated based on the AMD grade at the end of the clinical trial with follow-up time of 3 years. Progressors were those individuals with early or intermediate AMD at baseline who progressed to advanced AMD during follow-up, and individuals with advanced AMD in one eye at baseline who progressed to advanced AMD in both eyes

SECONDARY OUTCOMES:
Association between age and incident Advanced AMD | baseline
  controlling for age (70 years or older versus younger than 70)
Association between gender and incident Advanced AMD | baseline
Association between Baseline AMD grade and incident Advanced AMD | baseline
  Baseline AMD grade was deﬁned as AREDS category 1 in both eyes (essentially free of age-related macular abnormalities), category 2 in the worst eye (mild changes including multiple small drusen, nonextensive intermediate drusen, and/or pigment abnormalities), category 3 in the worst eye (at least one large drusen of at least 125µm diameter, extensive intermediate drusen, and/or noncentral geographic atrophy), category 4 in one eye (advanced AMD, either neovascular or central geographic atrophy, or visual loss due to AMD regardless of phenotype), or category 4 in both eyes.
Association between cigarette smoking and incident Advanced AMD | baseline
  cigarette smoking information was acquired by questionaires(never, past, or current)
  .
Association between body mass index (BMI) and incident Advanced AMD | baseline
  BMI was calculated as the weight in kilograms divided by the square of the height in meters ( 25, 25-29.9, and 30 )

CONTACTS AND LOCATIONS:
Overall Officials: Xiaoling Liu, MD, Principal Investigator — The Eye Hospital of Wenzhou Medical University
Locations (1):
- The eye hospital of Wenzhou Medical University, Wenzhou, Zhejiang, China

REFERENCES:
- [Background] Resnikoff S, Pascolini D, Etya'ale D, Kocur I, Pararajasegaram R, Pokharel GP, Mariotti SP. Global data on visual impairment in the year 2002. Bull World Health Organ. 2004 Nov;82(11):844-51. Epub 2004 Dec 14. PMID 15640920
- [Background] Huang EJ, Wu SH, Lai CH, Kuo CN, Wu PL, Chen CL, Chen CY, King YC, Wu PC. Prevalence and risk factors for age-related macular degeneration in the elderly Chinese population in south-western Taiwan: the Puzih eye study. Eye (Lond). 2014 Jun;28(6):705-14. doi: 10.1038/eye.2014.55. Epub 2014 Mar 14. PMID 24625378
- [Background] Ye H, Zhang Q, Liu X, Cai X, Yu W, Yu S, Wang T, Lu W, Li X, Jin H, Hu Y, Kang X, Zhao P. Prevalence of age-related macular degeneration in an elderly urban chinese population in China: the Jiangning Eye Study. Invest Ophthalmol Vis Sci. 2014 Sep 4;55(10):6374-80. doi: 10.1167/iovs.14-14899. PMID 25190650
- [Background] Mitchell P, Smith W, Attebo K, Wang JJ. Prevalence of age-related maculopathy in Australia. The Blue Mountains Eye Study. Ophthalmology. 1995 Oct;102(10):1450-60. doi: 10.1016/s0161-6420(95)30846-9. PMID 9097791
- [Background] Mitchell P, Wang JJ, Foran S, Smith W. Five-year incidence of age-related maculopathy lesions: the Blue Mountains Eye Study. Ophthalmology. 2002 Jun;109(6):1092-7. doi: 10.1016/s0161-6420(02)01055-2. PMID 12045049
- [Background] Yang K, Liang YB, Gao LQ, Peng Y, Shen R, Duan XR, Friedman DS, Sun LP, Mitchell P, Wang NL, Wong TY, Wang JJ. Prevalence of age-related macular degeneration in a rural Chinese population: the Handan Eye Study. Ophthalmology. 2011 Jul;118(7):1395-401. doi: 10.1016/j.ophtha.2010.12.030. Epub 2011 Mar 27. PMID 21444116
- [Background] Schmitz-Valckenberg S, Bultmann S, Dreyhaupt J, Bindewald A, Holz FG, Rohrschneider K. Fundus autofluorescence and fundus perimetry in the junctional zone of geographic atrophy in patients with age-related macular degeneration. Invest Ophthalmol Vis Sci. 2004 Dec;45(12):4470-6. doi: 10.1167/iovs.03-1311. PMID 15557456
- [Background] Johnson EJ, Chung HY, Caldarella SM, Snodderly DM. The influence of supplemental lutein and docosahexaenoic acid on serum, lipoproteins, and macular pigmentation. Am J Clin Nutr. 2008 May;87(5):1521-9. doi: 10.1093/ajcn/87.5.1521. PMID 18469279
- [Background] Tan JS, Wang JJ, Flood V, Rochtchina E, Smith W, Mitchell P. Dietary antioxidants and the long-term incidence of age-related macular degeneration: the Blue Mountains Eye Study. Ophthalmology. 2008 Feb;115(2):334-41. doi: 10.1016/j.ophtha.2007.03.083. Epub 2007 Jul 30. PMID 17664009
- [Background] Lovie-Kitchin J, Feigl B. Assessment of age-related maculopathy using subjective vision tests. Clin Exp Optom. 2005 Sep;88(5):292-303. doi: 10.1111/j.1444-0938.2005.tb06713.x. PMID 16255688
- [Background] Ying GS, Maguire MG, Alexander J, Martin RW, Antoszyk AN; Complications of Age-related Macular Degeneration Prevention Trial Research Group. Description of the Age-Related Eye Disease Study 9-step severity scale applied to participants in the Complications of Age-related Macular Degeneration Prevention Trial. Arch Ophthalmol. 2009 Sep;127(9):1147-51. doi: 10.1001/archophthalmol.2009.189. PMID 19752423